CLINICAL TRIAL: NCT06479122
Title: Efficacy of Intravenous Acetaminophen Alone Versus Combination of Acetaminophen/Ibuprofen (Maxigesic®IV) in Multimodal Analgesia After Cesarean Section: a Randomized Controlled Trial
Brief Title: Efficacy of Acetaminophen Alone Versus Combination of Acetaminophen/Ibuprofen After Cesarean Section
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2405-052-1535
Record Dates: First submitted 2024-06-18; First posted 2024-06-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cesarean Section; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen (Active Comparator)
  Interventions: Drug: Acetaminophen
- Acetaminophen/Ibuprofen (Experimental)
  Interventions: Drug: Acetaminophen/Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — 1g acetaminophen is administered during skin closure (end of operation).
  Other Names: Acetaminophen #1
  Arms: Acetaminophen
Drug: Acetaminophen/Ibuprofen — A mixture of 1g acetaminophen and 300 mg ibuprofen (Maxigesic®IV) is administered during skin closure (end of operation)
  Other Names: Acetaminophen/Ibuprofen #1
  Arms: Acetaminophen/Ibuprofen
Drug: Acetaminophen — 1g acetaminophen is administered 6 hours after the first administration.
  Other Names: Acetaminophen #2
  Arms: Acetaminophen
Drug: Acetaminophen/Ibuprofen — A mixture of 1g acetaminophen and 300 mg ibuprofen (Maxigesic®IV) is administered 6 hours after the first administration.
  Other Names: Acetaminophen/Ibuprofen #2
  Arms: Acetaminophen/Ibuprofen

SUMMARY:
The investigators aim to compare the analgesic efficacy of intravenous acetaminophen alone versus combination of acetaminophen/ibuprofen (Maxigesic®IV) in multimodal analgesia after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cesarean section
* Gestational age > 37+0 weeks

Exclusion Criteria:

* Emergency cesarean section
* Multiple pregnancy (e.g. twins, triplets)
* Body weight < 50 kg
* Preeclampsia
* History of hypersensitivity to acetaminophen or ibuprofen
* History of upper gastrointestinal tract bleeding or gastric ulcer
* Underlying liver disease
* Underlying kidney disease or GFR < 90 mL/min/1.73m2
* Heart failure or severe hypertension
* History of asthma
* Chronic use of barbital or tricyclic antidepressants

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Obstetric QoR-11K score 24 hours after end of surgery | 24 hours after end of surgery
  Minimum 0, poor recovery; maximum 110, good recovery

SECONDARY OUTCOMES:
Numeric rating scale pain score (0-10) 4 hours after end of surgery | 4 hours after end of surgery
  0, no pain; 10, worst pain imaginable
Numeric rating scale pain score (0-10) 8 hours after end of surgery | 8 hours after end of surgery
  0, no pain; 10, worst pain imaginable
Numeric rating scale pain score (0-10) 12 hours after end of surgery | 12 hours after end of surgery
  0, no pain; 10, worst pain imaginable
Numeric rating scale pain score (0-10) 24 h after end of surgery | 24 h after end of surgery
Numeric rating scale pain score (0-10) 48 hours after end of surgery | 48 hours after end of surgery
  0, no pain; 10, worst pain imaginable
Use of patient-controlled analgesia (FTN, micrograms) during the first 24 hours after end of surgery | 24 h after end of surgery
Use of patient-controlled analgesia (FTN, micrograms) during the first 48 hours after end of surgery | 48 h after end of surgery
Use of rescue analgesia during the first 24 hours after end of surgery | 24 h after end of surgery
Use of rescue analgesia during the first 48 hours after end of surgery | 48 h after end of surgery
Wound-related complications during hospital stay, up to 5 days | From end of surgery to patient discharge, up to 5 days
Operation time | Duration of operation
Anesthesia time | Duration of anesthesia
Injection level of intrathecal drug | After arrival at the operating room
Dosage of intrathecal drug (mg, bupivacaine) | After arrival at the operating room
Sensory blockade level by time point | 0, 5, 10 minutes after intrathecal injection and at the end of operation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided